CLINICAL TRIAL: NCT05777109
Title: A Dual-center, Randomized, Double-blinded and Parallel-controlled Study to Assess the Pharmacokinetic, Pharmacodynamics, Safety and Immunogenicity of HS-20090 Injection and Xgeva® in Healthy Adults
Brief Title: Comparing of the PK, PD, Safety and Immunogenicity of HS-20090 and Xgeva® in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HS-20090-102
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: HS-20090; Pharmacokinetic; pharmacodynamics; Safety; Immunogenicity
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-20090 (Experimental): Subcutaneously injection of HS-20090 (120mg/1.7mL) once on the first day
  Interventions: Drug: HS-20090
- Xgeva® (Active Comparator): Subcutaneously injection of Xgeva® (120mg/1.7mL) once on the first day
  Interventions: Drug: Xgeva®

INTERVENTIONS:
Drug: HS-20090 — A human IgG2 monoclonal antibody with affinity and specificity for human RANKL
  Other Names: Recombinant human anti-RANKL monoclonal antibody injection
  Arms: HS-20090
Drug: Xgeva® — Xgeva® injection (120mg) by subcutaneous injection once on the first day subcutaneous injection of 120 mg (1.7 ml)only once
  Other Names: Denosumab Injection
  Arms: Xgeva®

SUMMARY:
A Dual-center , Randomized, double-blinded and Parallel-controlled Study to Assess the Pharmacokinetic, pharmacodynamics, Safety and Immunogenicity of HS-20090 Injection and Xgeva® in Healthy Adults

DETAILED DESCRIPTION:
This is a phase I, dual-center, randomized, double-blind and parallel group clinical trial .

The primary objective is to assess the pharmacokinetic similarity of single subcutaneously injection of HS-20090 or Xgeva® in healthy volunteers.

The secondary objectives are to assess the Clinical safety and immunogenicity similarity of single subcutaneously injection of HS-20090 or Xgeva® in healthy volunteers. Meanwhile, observing the pharmacodynamic similarity of HS-20090 to Xgeva® preliminarily.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form and fully understand the test content, process and possible adverse reactions, and be able to complete the study according to the test plan requirements;
* Healthy males, Aged ≥18 years and ≤50 years old(including the boundary value);
* Subjects weighing ≥ 55 kg and ≤ 75 kg (weight difference in a single center is controlled within 10 kg), with a BMI between 19.0 and 26.0 kg/m2 (BMI = weight (kg)/height2 (m2)) (including borderline values).
* The subject agrees to use effective contraception for at least 6 months from the screening date until after study dosing, and has no plans to have children or donate sperm within 6 months;
* Physical examination, vital signs, laboratory examination, chest X-ray, B-ultrasound and electrocardiogram are normal, or the above tests are abnormal without clinically significance and have no effect on the test as judged by the investigator;
* ECG examination: corrected QT interval (QTcF) < 450 ms.

Exclusion Criteria:

* Occurred or suffering from osteomyelitis or ONJ (OsteoNecrosis of the Jaw) previously; The dental or jaw disease that is active, requiring oral surgery; or planned for invasive dental surgery during the study; or dental or oral surgery wounds have not healed;
* Subjects with any previous or current clinically serious diseases such as circulatory, endocrine, neurological, digestive, respiratory, genitourinary, hematological, immunological, psychiatric, and metabolic abnormalities or any other diseases that can interfere with the study results.
* Positive screening for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, Acquired Immune Deficiency Syndrome (AIDS) antibodies, and syphilis spirochete antibodies.
* Abnormal blood calcium: current hypocalcemia or hypercalcemia. Serum calcium outside the normal laboratory range; (Subjects should not apply calcium supplements for at least 8 hours prior to drawing blood for serum calcium screening assays.)
* previous use of RANKL inhibitors or osteoclastogenesis inhibitory factor.
* The subject is participating in another clinical study, or the first dose was administered less than 3 months after the last dose of the previous clinical study (or 5 half-lives of the study drug, whichever is longer).
* Average daily smoking ≥ 5 cigarettes in the 3 months prior to randomization.
* Prior history of alcohol abuse (14 units of alcohol per week: 1 unit = 360 mL of beer or 45 mL of spirits at 40% alcohol or 150 mL of wine), substance abuse or drug use.
* Positive substance abuse screening or/and alcohol breath test screening prior to study administration.
* Subjects who have donated blood within 3 months prior to administration, or have lost more than 400 ml of blood, or are scheduled to donate blood within 6 months.
* Subjects who have had a significant change in physical status within 6 months prior to administration, or who have been performing strenuous exercise.
* Subjects who, in the opinion of the investigator, have any factors that make participation in this trial inadvisable.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-04-05 (Estimated); Study Completion 2024-04-05 (Estimated)

PRIMARY OUTCOMES:
AUC0-∞ | 155days
  The area under the curve from time 0 extrapolated to infinite time
Cmax | 155days
  Maximum concentration

SECONDARY OUTCOMES:
AUC0-t | 155days
  Area under the plasma concentration-time curve
Tmax | 155days
  Time to reach Cmax
t1/2z | 155days
  Terminal half-life
Vz/F | 155days
  Apparent volume of distribution
CLz/F | 155days
  Apparent clearance
Serum type 1 C-telopeptide(CTX1) | 155days
  explore the pharmacodynamic profile by detecting the serum concentration of CTX1
Imin | 155days
  The minimum observed concentration
TEmax | 155days
  Time to reach the maximum inhibition rate
Emax | 155days
  Maximum observed inhibition rate
AUEC0-t | 155days
  Area under the plasma effect-time curve from time zero to last time of quantifiable concentrationthe
Adverse events(AE) | 155days
  The adverse medical events that occur after the clinical trial subjects receive the test drug do not necessarily have a causal relationship with the treatment.
Antidrug antibody(ADA): | 155days
  percentage of subjects positive for antidrug antibody
Neutralizing antibody(Nab) | 155days
  percentage of subjects positive for Nab

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoai He, Master, Principal Investigator — Haikou People's Hospital; Wei Zhao, Ph.D, Principal Investigator — Shandong First Medical University
Locations (1):
- Haikou People's Hospital, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No